CLINICAL TRIAL: NCT06137859
Title: Physical Literacy-based Intervention (PLBI) for Older Adults: A Cluster Randomized Controlled Trial Study Protocol
Brief Title: Physical Literacy-based Intervention for Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Sum Kim Wai Raymond, Dr, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBRE-21-0353
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Competence; Physical Activity; Knowledge, Attitudes, Practice; Motivation; Confidence, Self; Peer Group
Keywords: Physical literacy
MeSH Terms: conditions — Motor Activity; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive PLBI intervention treatment including weekly-based functional fitness training, mastering physical literacy class, daily based reflective writing, buddy peers support group.
  Interventions: Behavioral: Weekly-based functional fitness training; Behavioral: Mastering Physical Literacy Class; Behavioral: Daily based reflective writing; Behavioral: Buddy Peers Support Group
- Control (No Intervention): Participants will not receive PLBI intervention treatment. However, participants in the control group will be given the same treatment (program and activities) after all data has been collected.

INTERVENTIONS:
Behavioral: Weekly-based functional fitness training — Participants will receive a 12-week duration of functional fitness training in daycare centers, which will be implemented twice a week. The 60-minute per session training series will be delivered and guided by qualified elderly health and fitness instructors, who will be provided with a workshop before this intervention. The workshop will be designed and delivered by the research team. The first session will focus on the physical literacy of older adults and the second session will focus on how to lead functional fitness training under the FITT principle for older adults. The main goal of functional training is to improve the range of joint motion, increase muscle strength and flexibility, and boost blood circulation safely. Therefore, symmetry training together with cardiovascular training is the core of the training program. Examples of the main training activities include cardio-full-body exercises, upper-body exercises, lower-body exercises and sensory integrative training.
  Arms: Intervention
Behavioral: Mastering Physical Literacy Class — A 30-minute MPLC program will be conducted by experienced elderly health and fitness instructors after WBFFT. This MPLC program aims to enhance the knowledge and understanding of physical literacy. Referring to the newly developed consensus statement, the MPLC includes the following five domains related to the relationship with movement and physical activity throughout life:
  i) Why physical literacy matters - improves health, well-being and quality of life.
  ii) Understanding physical literacy - value, enjoy and engage in physical activity for life.
  iii) Everyone's physical literacy is different - their individual needs and experiences of movement and physical activity.
  iv) Building physical literacy - think, feel, move and connect with others. v) How experience affects physical literacy - people, places and spaces around us.
  Arms: Intervention
Behavioral: Daily based reflective writing — At the end of the baseline stage of this study, each participant of the intervention group will receive a template notebook for daily-based reflective writing. The required columns consist of the daily diet, physical activity, mood and sleep quality. Participants will be required to write down their behavior in this notebook daily. In each week's functional training course, there will be a life-sharing session, where the participants will be reminded to bring their notebooks and share their daily activities with others. They will receive feedback, advice and encouragement from the instructor and each other. The notebook will be collected during the last week of the intervention.
  Arms: Intervention
Behavioral: Buddy Peers Support Group — Peer-support groups with buddy members will be arranged in each daycare center. Three pairs of buddies and hence about 6 participants will be formed per group. A total of 6 buddy pairs and 2 groups will be formed per daycare center. Buddy peers will encourage each other to do functional exercises regularly or to perform functional exercises together. The time and place for the practice will be decided among buddy members. A member in each group will be nominated as the leader to assist in the liaison and coordination of group activities. The group will perform weekly group-based functional exercises, and the time and place for the practice will be decided among group members. The group will be encouraged to hold monthly gatherings with their fitness instructor in order to strengthen social support.
  Arms: Intervention

SUMMARY:
The ageing population creates concerns and challenges worldwide. The large number of older adults (aged over 65) in Hong Kong continues to rise as people live longer. This may result in heavy burdens on public services and problems such as a shortage of medical resources.

The purpose of this study is to implement a physical literacy-based intervention (PLBI) among older adults in Hong Kong in order to achieve the goal of health promotion. A two-arm cluster randomized controlled trial will be employed in this proposed study. Ten daycare centers for the elderly in Hong Kong will be invited to participate in this study. The intervention group will receive functional fitness training and mastering physical literacy class twice a week with buddy peer support, and they will be asked to keep a reflective writing journal on a daily basis for 12 weeks in total. Participants will be evaluated at baseline (week 0), post-intervention (week 12), and at 6-week follow-up (week 18). This will consist of objective and self-reported measures covering elements within physical literacy (i.e. physical competence, motivation and confidence, knowledge and understanding) and also physical activity levels on an individual basis.

The study intends to introduce a conceptual framework of physical literacy for the elderly through an intervention that allows older people to develop daily behaviour habits, which should promote active ageing for the elderly and greater self-esteem in later life. After this study, participants may share their positive experiences, and encourage their peers in the community to become physically literate in the future. In the long run, due to the feasibility and sustainability of these potential programs, this proposed study has the potential to connect seniors through social engagement and contribute to healthy living.

DETAILED DESCRIPTION:
Older adults who are physically literate can effectively adapt to physical challenges associated with injury, chronic disease, and aging, demonstrating a characteristic ability to maintain their independence for an extended period compared to those who engage in less physical activity. Older adults who are physically literate can adapt to challenges associated with injury, chronic disease, and aging, thereby maintaining their independence for a more extended period compared to those who engage in less physical activity. Viewed through the lens of physical literacy, successful agers adeptly adjust and modify their activities, employing age adaptation and physical competence. They achieve this by optimizing their choices in terms of motivation and enjoyment of movement, ultimately maximizing their success, boosting confidence, and sustaining higher levels of functioning across all dimensions. Thus, developing physical literacy aligns with the goal of promoting healthy ageing, enhancing the prospects for overall well-being across the lifespan. This is grounded in the understanding that initiating an active lifestyle from the outset contributes to preserving independence and positively impacting population health.

This study attempts to introduce a conceptual framework of physical literacy through a Physical Literacy Based Intervention (PLBI) that allows older adults to develop good exercise habits with the development of daily behavioral habits. Based on the unique physical literacy journey and lifestyle of each individual, the proposed study would offer the elderly a meaningful way to achieve active ageing and encourage them to realize their physical literacy journey in later life. Evidence has shown that exercise is associated with better physical and mental health in older adults, and exercising with others is more likely to lead to a sufficient amount of physical activity. After this study, it is expected that older people will also encourage their peers in the community to engage in physical activity.

The benefits of physical activity to health are widely acknowledged. The concept of physical literacy has been vaunted as a key component in the establishment of lifelong adherence to physical activity. McLennan and Thompson espouse that physical literacy is the foundation of quality physical education. The development of physical literacy is the most influential variable with respect to physical health improvement. The proposed research, therefore, aims to implement a PLBI including functional fitness training and mastering physical literacy class, buddy peer support, and reflective writing for the development of motivation, confidence, physical competence, knowledge and understanding under the concept of physical literacy to achieve the goal of health promotion. This will add an effective comprehensive assessment and charting of physical literacy for older adults. In the short term, this study will lead to a convenient and powerful program and assessment tool that can be used by elderly centers and elderly fitness trainers and assessors. In the long term, this research will benefit the general public, in particular, communities of older people by encouraging participation in physical activity. When framing the proposed model to chart physical literacy for older adults, the program and measurement system may be adopted in elderly and ageing studies.

The aims of this study are 1) to develop and implement a PLBI including functional fitness training, mastering physical literacy class, buddy peers support, and reflective writing for older adults in Hong Kong; 2) to explore physical literacy (physical competency, daily behavior, knowledge and understanding, and motivation and confidence) of the older adults in Hong Kong; 3) to examine the effectiveness of a PLBI in terms of changes in physical literacy development among older adults in Hong Kong; and 4) to add information to the literature of physical literacy, gerontology, and public health in the Asian context of Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* those aged 65 to 74 years old who are registered in a daycare center/unit for the elderly in Hong Kong.
* the ability to walk eight meters without assistance.
* able to read and write.

Exclusion Criteria:

* neurological disease which impairs mobility, cardiovascular disease which results in shortness of breath or angina on walking up one flight of stairs.
* cognitive impairment. Participants' cognitive function will be screened by the Chinese Mini-Mental State Examination and those who score below 24 will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Competence | Week 0; Week 12; Week 18
  Short Physical Performance Battery (SPPB) will be used to measure the physical competence within the physical literacy of older adults. Huang et al. suggested using a combined and comprehensive kit of assessment tools to measure physical competence, and the SPPB was reported to be able to measure complex capabilities with excellent test-retest reliability, especially in community-dwelling older adults. It is a group of measures that combines the results of the gait speed, chair stand and balance tests, which consist of balance, a timed eight feet walk and chair stands. The scores range from zero (worst performance) to 12 (best performance). It has been used as a predictive tool for possible disability and can aid in monitoring function in older people. The reliability of SPPB has been reported as ICC = 0.75 - 0.89 for all measures.
Objective Physical activity levels | Week 0; Week 12; Week 18
  Accelerometers (Actigraph wGT3X-BT) will be used to measure the physical activity engagement levels of participants, and are categorized as sedentary, light, moderate and vigorous. Data was collected in 60 s epochs to account for elderly people's natural activity levels, as it was shown to present the most acceptable classification accuracy for accelerometer use among older adults. The cut-points developed by Aguilar-Farías et al. was applied to identifying intensity levels. Participants will wear accelerometers at the waist to measure their physical activity engagement levels for at least 8 hours per day, for seven consecutive days.

SECONDARY OUTCOMES:
Demographic information | Week 0; Week 12; Week 18
  Demographic information including age, gender, BMI (heigh and weight), education, and socio-economic status will be included in the starting part of the questionnaire set, in order to acquire personal characteristics for further analysis.
Self-report physical activity levels | Week 0; Week 12; Week 18
  International Physical Activity Questionnaire - short form is the short version of the International Physical Activity Questionnaire used to measure self-reported physical activity levels. They will be required to report on the total duration of different types of physical activity which lasted at least 10 uninterrupted minutes in the last 7 days. Example item included: During the last 7 days, how many days did you do vigorous physical activities?
Knowledge and understanding | Week 0; Week 12; Week 18
  Montreal Cognitive Assessment (MoCA) is a 30-question brief and sensitive test used for detecting Alzheimer's disease and measuring executive functions and multiple cognitive domains. It is widely adopted for older adults and will be used to assess knowledge and understanding of physical literacy among the elderly. MoCA-B is a revised MoCA test. The Chinese Version of MoCA-B tests nine cognitive domains (executive function, language, orientation, calculation, conceptual thinking, memory, visual perception, attention, and concentration), and has been reported as a reliable cognitive screening test across all education levels in Chinese elderly adults, with high acceptance and good reliability.
Physical literacy | Week 0; Week 12; Week 18
  Perceived Physical Literacy Instrument (PPLI) is a 9-item instrument which is used to measure the perceived physical literacy of different individuals. Three sub-scales are "sense of self and self-confidence", "self-expression and communication with others" and "knowledge and understanding" which were identified as key attributes of physical literacy (4). Participants responded to the instrument on a 1 to 5 Likert scale (1 = strongly disagree and 5 = strongly agree). Sum et al. confirmed that the three-factor validity (RMSEA = 0.08; CFI = 0.94 and SRMR = 0.04) and convergent validity (CR = 0.72 - 0.78; AVE = 0.43 - 0.54) of the PPLI was satisfactory.
Motivation and confidence | Week 0; Week 12; Week 18
  Perceived Well-being Scale (PWB) contains 14 items with 7 points which will be used to measure participants' motivation and confidence. It is a short and convenient measure for use with community-based and institutionalized elderly. Example items include: (a) I am often bored (psychological well-being); (b) I am in good shape physically (physical well-being). The validity of PWB is sufficiently high to justify being used with the elderly, in particular in longitudinal and intervention studies.
Buddy Peers Support | Week 0; Week 12; Week 18
  A 5-item Friend Support for Exercise Habit Subscale of the validated Social Support for Diet and Exercise Behavior Scale will be used. Five questions are "exercise with me", "offered to exercise with me", "gave me reminder to exercise", "gave me encouragement to stick with my exercise program", and "changed their schedule so we could exercise together". Participants responded to the instrument on a 1 (none) to 5 (very often) Likert scale. Sallis et al. confirmed that the sub-scales are with high acceptance and good reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Wai Raymond Sum, EdD, Principal Investigator — Chinese University of Hong Kong

REFERENCES:
- [Derived] Sum RKW, Yang Y, Choi SM, Duncan MJ, Li M. Physical literacy-based intervention for older adults: a cluster randomized controlled trial study protocol. Front Sports Act Living. 2024 Jul 17;6:1392270. doi: 10.3389/fspor.2024.1392270. eCollection 2024. PMID 39086857

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT06137859/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT06137859/ICF_001.pdf